CLINICAL TRIAL: NCT01622647
Title: The Effect of Nasal Continuous Positive Airway Pressure (N-CPAP) on Arterial pCO2 During Spinal Anesthesia With Intravenous Sedation for Total Knee Arthroplasty
Brief Title: The Effect of Nasal Continuous Positive Airway Pressure (N-CPAP) on Arterial pCO2 During Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatrix (Other)
Collaborators: New Hanover Regional Medical Center (Other); American Anesthesiology of the Carolinas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-Z078-1611
Record Dates: First submitted 2012-06-05; First posted 2012-06-19 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Knee Replacement Surgery
Keywords: NCPAP
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NCPAP Group (Active Comparator): Group of patients that do receive NCPAP treatment
  Interventions: Other: Nasal Continuous Positive Airway Pressure (NCPAP)
- No NCPAP (No Intervention): subjects will not receive NCPAP

INTERVENTIONS:
Other: Nasal Continuous Positive Airway Pressure (NCPAP) — Subjects will receive NCPAP
  Arms: NCPAP Group

SUMMARY:
The proposed study intends to investigate several aspects of the respiratory effects of intravenous sedation of patients undergoing spinal anesthesia for knee replacement surgery. The study will include assessment of PaCO2 during the intraoperative period. PaCO2 is expected to be elevated as a result of intravenous sedation and postural factors. Further, the study will investigate how application of Nasal Continuous Positive Airway Pressure (N-CPAP) may impact PaCO2.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology Class I, II, or III patients
* Age over 21 years and under 70 years
* Planned surgical procedure is total knee arthroplasty (TKA) to be performed at Cape Fear Hospital
* Body Mass Index less than 40
* The patient and their attending anesthesiologist select spinal anesthesia with intravenous sedation, intrathecal morphine, and femoral nerve block as the preferred anesthesia plan

Exclusion Criteria:

* Prior diagnosis of Obstructive Sleep Apnea based upon sleep study
* History of Stroke with residual neurologic deficit
* Prior diagnosis of Emphysema, Chronic Bronchitis, Chronic Obstructive Pulmonary Disease, or Asthma, or other chronic lung disease
* Recent history of significant nasal obstruction, epistaxis, or facial abnormality that may interfere with proper fit of a nasal CPAP mask
* Pregnancy
* Mental or other disability preventing a patient from personally giving informed consent
* Chronic narcotic or benzodiazepine treatment or dependency
* Allergy to Midazolam, Fentanyl, or Propofol
* Severe upper respiratory infection within the past three weeks

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Arterial Blood Gas (ABG) test to investigate the breathing effects on patients receiving CPAP treatment during spinal anesthesia for knee replacement. | ABG will be collected five minutes after surgical skin incision and the second specimen will be collected exactly 30 minutes later.
  The TEST patients will receive CPAP treatment immediately after the first ABG specimen is drawn. After collection of the second ABG specimen, the anesthesia team may elect to remove the N-CPAP mask or maintain it as deemed best. The CONTROL patients will not receive CPAP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Smith, MD, Principal Investigator — American Anesthesiology of the Carolinas
Locations (1):
- New Hanover Regional Medical Center, Wilmington, North Carolina, United States